CLINICAL TRIAL: NCT05940545
Title: UMIT-1 Trial: Favipiravir & Ribavirin Phase IB A Randomised Phase Ib Study to Determine the Phase II Dose and to Evaluate the Safety and Efficacy of Intravenous (IV) Favipiravir & Ribavirin
Brief Title: UMIT-1 Trial Favipiravir & Ribavirin for the Treatment of CCHF
Acronym: UMIT-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-021
Record Dates: First submitted 2023-05-03; First posted 2023-07-11 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-06

CONDITIONS: CCHF
MeSH Terms: interventions — favipiravir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 (Active Comparator): 6 patients will be randomised to starting dose of favipiravir 1800 mg BD (day 1), then 800mg BD Day 2 to 10, or standard of care.
  Interventions: Drug: Favipiravir
- Cohort 2 (Active Comparator): 6 patients will be randomised to starting dose of favipiravir 2600 mg BD (day 1), then 1200mg BD day 2 to 10, or standard of care.
  Interventions: Drug: Favipiravir
- Cohort 3 (Active Comparator): 6 patients will be randomised to starting dose of favipiravir 1800 mg BD (day 1), then 800mg BD Day 2 to 10 plus Ribavirin, or standard of care.
  Interventions: Drug: Favipiravir; Drug: Ribavirin
- Cohort 4 (Active Comparator): 6 patients will be randomised to starting dose of favipiravir 2600mg BD (day 1), then 1200mg BD day 2 to 10 plus Ribavirin, or standard of care.
  Interventions: Drug: Favipiravir; Drug: Ribavirin

INTERVENTIONS:
Drug: Favipiravir — Small molecule antiviral
Drug: Ribavirin — Small molecule antiviral
  Arms: Cohort 3; Cohort 4

SUMMARY:
UMIT-1: A Randomised Phase Ib Study to Determine the Phase II dose and to Evaluate the Safety and Efficacy of intravenous (IV) Favipiravir & Ribavirin for the Treatment of CCHF

DETAILED DESCRIPTION:
This will be a 2:1 randomised open-label phase I trial of IV Favipiravir and IV Favipiravir plus Ribavirin vs optimised standard of care in CCHF. The phase Ib will be carried out to test the safety and tolerability of IV Favipiravir in hospitalised patients. Following review of safety, tolerability and PK data from evaluated phase I doses, an IV Favipiravir doses will be selected to progress to phase II. virological efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult in-patients (≥18 years) with laboratory confirmed CCHF infection by positive polymerase chain reaction (PCR) test.
2. Ability to provide informed consent signed by study patient or legally acceptable representative
3. Women of childbearing potential (WOCBP) and male patients who are sexually active with WOCBP must agree to use a highly effective method of contraception (as outlined in section 5.4 below) from the first administration of trial treatment, throughout trial treatment and for the duration outlined in trial protocol as well as addition 14 days for women and 7 days for men after the last dose of trial treatment.
4. Severity Grading System (SGS) for CCHF - mild/moderate.
5. Less than or equal to 7 days from onset of CCHF symptoms

Exclusion Criteria:

1. Stage 4 severe chronic kidney disease or requiring dialysis (i.e., estimated glomerular filtration (eGFR) rate <30 mL/min/1.73 m2)
2. Pregnant or breast feeding
3. Anticipated transfer to another hospital which is not a study site within 72 hours
4. Known Allergy to any study medication
5. Patients participating in another clinical trial of an investigational medicinal product (CTIMP) within the last 30 days.
6. Positive COVID-19 PCR
7. Previous intolerance of Favipiravir or Ribavirin
8. Haemoglobinopathies
9. Unstable cardiac diseases within 6 months
10. Any participants deemed not suitable, based on investigators opinion.
11. Patients taking the drugs listed in section 8.11 within 30 days or 5 times the half-life (whichever is longer) of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety objective To determine the safety and tolerability of multiple doses of IV Favipiravir in patients with CCHF | Up to day 8
  Adverse events and serious adverse events
  Dose limiting toxicities (Safety and Tolerability of IV Favipiravir and IV Favipiravir/Ribavirin- CTCAE v5 Grade ≥3 adverse events)
To determine the safety and tolerability of multiple doses of IV Favipiravir in combination with Ribavirin in patients with CCHF | up to day 8
  Adverse events and serious adverse events
  Dose limiting toxicities (Safety and Tolerability of IV Favipiravir and IV Favipiravir/Ribavirin- CTCAE v5 Grade ≥3 adverse events)

SECONDARY OUTCOMES:
Pharmacokinetic objective: To characterise the plasma pharmacokinetics of multiple doses of IV Favipiravir and IV Favipiravir in combination with Ribavirin | up to Day 8
  Evaluation of favipiravir in VHFs is limited by the predicted high-pill burden (up to 30 tablets per day) required and uncertainty around dose and PK.
  Favipiravir injection (IV favipiravir) is a novel formulation of favipiravir for intravenous drip infusion, with Cmax levels 4-fold higher following administration of multiple doses in cynomolgus monkeys compared to oral (Toyama IB).
  The favipiravir activity is derived from the intracellular ribofuranosyl-5'-triphosphate (RTP) metabolite that has a longer half-life intracellularly than the parent drug in plasma. Therefore, transiently higher Cmax values are expected to translate into sustained higher intracellular RTP concentrations and thus activity.
Virologic objective | Change from baseline over time, up to Day 29, in viral load
  To investigate the effect of IV Favipiravir alone and in combination with Ribavirin on CCHF viral load
Clinical objective | Mortality at Days 15 and 29
  To investigate the ability of IV Favipiravir and in combination with Ribavirin to reduce the duration of signs and symptoms of CCHF in-patients.
Clinical objective | Time from randomisation to death (up to day 29)
  To investigate the ability of IV Favipiravir and in combination with Ribavirin to reduce the duration of signs and symptoms of CCHF in-patients.

OTHER OUTCOMES:
Pharmacokinetic objective: To investigate the exposure-response relationship of IV Favipiravir on CCHF viral dynamics. | At End of study (6 Months)
  Change in host immune response
Pharmacokinetic objective: To investigate the exposure-response relationship of IV Favipiravir on CCHF viral dynamics. | At End of study (6 Months)
  Change in CCHFV culture and sequencing
Pharmacokinetic objective: To characterise virus and host immune response. | At End of study (6 Months)
  Change in host immune response
Pharmacokinetic objective: To characterise virus and host immune response. | At End of study (6 Months)
  Change in CCHFV culture and sequencing
Measure immune response by aldehyde oxidase (AO) / xanthine oxidase (XO) activity. | At End of study (6 Months)
  To investigate the exposure-response relationship of IV Favipiravir and IV Favirpiravir/Ribavirin on CCHF viral dynamics
  (Favipiravir inhibits AO and XO is partially involved in metabolism of favipiravir)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy E Read, PhD, MRCP, Study Director — Liverpool School of Tropical Medicine
Locations (1):
- Ankara Oncology Training and Research Center, Ankara, Yenimahalle, Turkey (Türkiye)